CLINICAL TRIAL: NCT01782846
Title: Double Blind-randomized Study Comparing the Efficacy of Two Analgesia (Ixprim® and Dafalgan-Codeine®) , in the Emergency Unit.
Brief Title: Trama-Code (Two Analgesics-comparative Study)
Acronym: Trama-Code
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010/45
Record Dates: First submitted 2013-01-25; First posted 2013-02-04 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Ixprim® (Active Comparator): 2 capsules of Ixprim® given orally (1000 mg Paracetamol + 75 mg Tramadol)
  Interventions: Drug: Ixprim®
- Dafalgan Codeine® (Active Comparator): Two capsules of Dafalgan Codeine® given orally (1000 mg Paracetamol + 46.8 mg Codeine)
  Interventions: Drug: Dafalgan-Codeine®

INTERVENTIONS:
Drug: Ixprim®
  Arms: Ixprim®
Drug: Dafalgan-Codeine®
  Arms: Dafalgan Codeine®

SUMMARY:
Double-blind randomized study to compare the efficacy of two analgesic drugs(Ixprim®, Dafalgan-Codeine®) in the emergency unit.

The efficacy (relief of pain) would be assessed 2 hours after administration of one of the two drugs in a patient presented to the emergency unit with a moderate pain (4 to 6 on pain assessment score).

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 - 75 years of age
* Presented to the emergency unit of FOCH hospital
* Complaining of moderate pain (4-6 on pain assessment scale) evaluated by the reception nurse

Exclusion Criteria:

* Patient already had received another type 2 analgesia or already received one of the study drugs in the last 4 hours
* pregnant or lactating females
* Patient with one or more contraindication to one of the study drugs
* Patients for whom the pain assessment scale can not be performed (unconscious, confused ...)
* Patient cannot be included for legal reasons
* Patient required urgent management
* Patient for whom it is considered difficult to be reassessed 2 hours later
* Patient unable to swallow

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
pain improvement | 120 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital FOCH - Emergency unit, Suresnes, Île-de-France Region, France